CLINICAL TRIAL: NCT05335681
Title: Midwife Öznur Hayat Öktem
Brief Title: The Effects of Warm Showers Application in Birth on Birth Pain, Birth Satisfaction and Birth Results
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Öznur Hayat Öktem, Midwife, principal investigator, Gulhane School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Hayat01; PhD midwifery (Registry Identifier: GulhaneSM)
Record Dates: First submitted 2022-04-02; First posted 2022-04-19 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Labor; Pregnancy; First Stage of Labor
Keywords: warm shower; labor pain; birth Satisfaction; hydrotherapy; maternal health
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: randomized controlled
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Warm Showers Application (Experimental): In the experimental group, a 20-minute warm shower (37 °C) will be administered when cervical dilation reaches at least 4 cm and again at 7 cm. The control group will receive standard care only. The hot shower will be applied to the sacral area, lower abdomen, and groin regions.
  Interventions: Behavioral: Warm Showers Application
- Standard Intrapartum Care (No Intervention): No intervention will be provided to the control group. At the stages when cervical dilation reaches 4 cm and 7 cm, pain will be evaluated using the VAS at baseline, 10 and 20 minutes.

INTERVENTIONS:
Behavioral: Warm Showers Application — In the experimental group, a 20-minute warm showers (37 °C) will be administered when cervical dilation reaches at least 4 cm and again at 7 cm. The control group will receive standard care only. The warm showers will be applied to the sacral area, lower abdomen, and groin regions.
  Throughout the intervention, the researcher will accompany the pregnant women to ensure safety and proper implementation of the procedure.
  Pain will be assessed using the VAS scale before the intervention and at 10 and 20 minutes after the intervention. The Birth Satisfaction Scale will be administered prior to discharge
  Arms: Warm Showers Application

SUMMARY:
The use of non-pharmacological methods in labor pain is very important in order to improve the birth process, increase comfort and provide relaxation. The role of midwives, acting as patient advocate is to maintain comfort throughout the birth process. In order to do this, she should know very well the non-pharmacological methods to be applied to the pregnant woman and choose the most appropriate one. Applying a warm shower, which is one of the non-pharmacological methods; the uterus Increases perfusion, makes labor painless felt, increases the release of oxytocin, and decreases the release of stress hormones.

In addition, while reducing the intervention rates, it improves birth and newborn outcomes and affects positively. Purpose of the research; labor pain of warm shower application, labor to evaluate the effect on satisfaction and birth outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 35,
* Having a singleton fetus between 37-42 weeks of gestation,
* Planning a a spontaneous vaginal birth,
* Having a cervical dilatation <5 cm.
* Having a fetus weighing between 2500-4000 grams,

Exclusion Criteria:

* Being short (<145cm),
* Being obese (BMI >30),
* Receiving pharmacological or non-pharmacological intervention for labor pain,
* Having chronic diseases during pregnancy (gestational diabetes, hypertension, preeclampsia,
* Undergoing operative vaginal delivery (forceps, vacuum),
* Making an emergency cesarean decision,
* Experiencing abnormal changes in fetal heart rates.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women who applied to the hospital for delivery
Enrollment: 78 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Labor Pain | Baseline (Before the cervical dilation)
  Visual analog scale:On a 10 cm (100 mm.) ruler, which is marked painlessness on one end and the most severe pain possible on the other, the patient expresses his or her own pain by drawing a line, pointing or pointing. The length of the distance from the point where there is no pain to the point marked by the patient is measured in centimeters and the numerical value found shows the severity of the patient's pain.
Labor pain | 10 minutes after the cervical dilation
  Visual analog scale.On a 10 cm (100 mm.) ruler, which is marked painlessness on one end and the most severe pain possible on the other, the patient expresses his or her own pain by drawing a line, pointing or pointing. The length of the distance from the point where there is no pain to the point marked by the patient is measured in centimeters and the numerical value found shows the severity of the patient's pain.
Labor pain | 20 minutes after the cervical dilation
  Visual analog scale.On a 10 cm (100 mm.) ruler, which is marked painlessness on one end and the most severe pain possible on the other, the patient expresses his or her own pain by drawing a line, pointing or pointing. The length of the distance from the point where there is no pain to the point marked by the patient is measured in centimeters and the numerical value found shows the severity of the patient's pain.

SECONDARY OUTCOMES:
Birth satisfaction | Pregnant women in both groups will be visited by the researcher in the postpartum service within the first 24 hours postpartum and BSC will be applied.
  The birth satisfaction scale (BSS).The scale is likert type and is scored as Strongly agree:5, Agree:4, Undecided:3, Disagree:2, Strongly disagree:1. Items 4, 8, 12, 15, 16, 17, 19, 20, 21, 23, 25, 29 are scored in reverse on the scale. The original form of the scale consists of 30 items, and the score that can be obtained from the scale varies between 30-150 points. As the score obtained from the scale increases, the satisfaction with the birth increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Öznur Hayat Öktem, Karabük, Turkey (Türkiye)